CLINICAL TRIAL: NCT00281073
Title: A Sequential Phase I - Phase II Pilot Study to Compare Cardiac Imaging Capabilities of ICE With TEE Followed by a Randomized Comparison of ICE Guided Cardioversion With Conventional Cardioversion Strategy in Patients With Atrial Fibrillation
Brief Title: Intra-Cardiac Echocardiography Guided Cardioversion(ICE-CHIP) Study
Acronym: ICE-CHIP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EP MedSystems (Industry)
Responsible Party: Sanjeev Saksena MD, Electrophysiology Research Foundation, Warren, NJ
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-01
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Atrial Fibrillation
Keywords: Intra-Cardiac Echocardiography; Cardioversion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TEE and ICE (Active Comparator): Serial use of TEE and ICE for comparative analysis
  Interventions: Device: Intra-Cardiac Echocardiography guided Cardioversion; Device: Intracardiac Echo; Device: ICE
- ICE or TEE (Active Comparator)
  Interventions: Device: ICE

INTERVENTIONS:
Device: Intra-Cardiac Echocardiography guided Cardioversion — Intracardiac Echo and TEE
  Arms: TEE and ICE
Device: Intracardiac Echo — Intracardiac Echo Viewmate
  Arms: TEE and ICE
Device: ICE — ICE or TEE

SUMMARY:
This is a sequential phase 1 and phase 2 study to evaluate the efficacy of intracardiac echocardiography to detect septal and left atrial pathology as compared to transesophageal echocardiography (Phase 1) and its value in a management strategy for immediate cardioversion during cardiac catheterization procedures in patients with atrial fibrillation as compared to a conventional strategy delaying cardioversion till full anticoagulation is established for a three weeks (Phase 2). Phase 1 will enroll 100 patients at 12 centers; these patients will be undergoing clinically indicated TEE & cardiac catheterization procedures. After review of Phase 1 results by an independent DSMB & the investigators that establish efficacy of ICE, Phase 2 will be initiated. Phase 2 will enroll 300 patients in 15 centers; these patients with atrial fibrillation will be undergoing clinically indicated cardiac catheterization procedures and have a clinical indication for cardioversion. Patients will be randomized to ICE guided cardioversion strategy or a conventional strategy employing three weeks of full anticoagulation before cardioversion. ICE imaging will be used to identify a low risk group for immediate cardioversion. A composite primary study endpoint that will include mortality and major morbidity including stroke and bleeding complications will be used.

This study will examines two hypotheses in AF patients undergoing invasive cardiac procedures:

Hypothesis 1: That ICE has comparable efficacy to TEE in visualization of left atrial pathology or septal defects that can predispose patients to stroke. This will be evaluated during the Phase I component of the study.

Hypothesis 2: That ICE can identify low risk patients in whom immediate cardioversion during the procedure is safe and comparably effective to electrical cardioversion performed based on a conventional strategy of a minimum of 3 weeks of preceding anticoagulation therapy. Low risk patients are expected to have an acceptably low incidence rate of stroke, transient ischemic attack (TIA), peripheral embolism, and major hemorrhagic events following electrical cardioversion. This will be evaluated during the Phase II component of the study, after the Phase I objective is achieved.

DETAILED DESCRIPTION:
The presence of intra-atrial thrombi or their precursors with their propensity for systemic embolism or the presence of interatrial septal defects are major concerns for patients with atrial fibrillation (AF) undergoing cardioversion. Transesophageal echocardiography (TEE) has been demonstrated to be a sensitive tool to detect septal defects, left atrial thrombi and spontaneous echo contrast (1, 2,3). The ACUTE trial documented that TEE based exclusion of intra cardiac thrombi, smoke or spontaneous echo contrast can facilitate safe immediate cardioversion in patients with AF. (4) This trial demonstrated comparable risk of embolic events with a TEE- based strategy to identify low risk patients for immediate cardioversion when compared to a conventional strategy of 3 weeks of anticoagulation before cardioversion.

The recognition of systemic thromboembolism as a significant potential complication of cardioversion during interventional cardiology procedures in patients with AF has stimulated interest in the clinical evaluation of catheter based intra cardiac echocardiography (ICE). Initial experience with intra cardiac phased -array imaging has demonstrated the efficacy and feasibility of this technology for intracardiac application and its capability in high resolution imaging of endocardial structures. (5) In the recent times, the utility of this imaging modality in various interventional procedures has been investigated and its effectiveness in visualizing left atrial thrombi during ablative procedures has been demonstrated in observational studies. (6 -11) However, a prospective multicenter comparative study of these two imaging techniques is unavailable. Should ICE provide comparable imaging capabilities to TEE, the value of ICE guided cardioversion during invasive procedures can also then be systematically studied during a prospective multicenter clinical study.

The ICE CHIP study is a prospective open label randomized multi-center investigation performed in two phases designed to initially compare two distinct imaging modalities (Phase 1) and subsequently two different strategies (ICE guided Cardioversion and Conventional) in the management of AF in patients undergoing invasive cardiac procedures in whom electrical cardioversion is indicated (Phase 2).

In Phase I, each patient will be imaged by TEE & ICE and a core echo laboratory will perform a blinded comparison of the two imaging modalities.

In Phase II, patients will be randomized to one of the two treatment groups. Investigators will be blinded to the method of management for each patient prior to their enrollment into the study. The composite incidence rate of major cardiac and bleeding complications (stroke, TIA, peripheral embolism, major hemorrhagic event) will be compared between the two treatment groups over the duration of the study.

In Phase 1, 100 patients will be enrolled at up to 12 investigational centers in USA & Europe. Study patients will have clinically indicated a TEE procedure as well as an invasive cardiac procedure. Recordings from both imaging methods will be analyzed in an independent and blinded manner at the core laboratory. It is estimated that enrollment will take 3 months.

In Phase 2, a total of 300 patients (3:2 randomization) will be enrolled in the study at up to 15 investigational sites in USA and Europe. Patients with AF who require electrical cardioversion will be enrolled into the study. The study will last for 8 weeks for each subject, with an estimated overall duration of 12 months (8 months enrollment period, 2 months follow-up period, remaining time for close-out) for the study.

The pilot study design was selected in order to evaluate the comparative accuracy of ICE imaging and TEE as well as the feasibility of ICE guided management of AF. In Phase 1, the design will ensure that ICE imaging is not inferior to standard TEE for detection of left atrial pathology. In Phase 2, ICE imaging will be performed in patients prior to immediate electrical cardioversion to determine if it is equivalent to the conventional management strategy of electrical cardioversion after anticoagulation for 3 weeks prior to cardioversion.

Both the Phase I and Phase II studies will be open label. An open label study design is proposed because it is not possible to blind the clinicians, patients or the sponsor to the identity of the diagnostic technique in Phase I (ICE vs. TEE) and to management strategy in Phase II (ICE vs. Conventional Strategy). The ICE and TEE data analysis in the Phase I component by the core lab will be blinded in so far as the identity of the patient, investigator and center. In the Phase II study, patient randomization to the treatment groups will minimize the chance of patient selection bias. An 8-week study duration was chosen for the Phase II component because most major cardiac and bleeding complications occur within this period.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the Phase I Component

1. Patients with spontaneous AF
2. Patients with or without structural Heart Disease.
3. Men or Women aged 18 years or older.
4. Patients undergoing an invasive catheterization procedure including right heart catheterization.
5. Patients who give an informed consent for participation in the study.
6. Patients who have undergone a trans-thoracic echocardiogram within the last 14 days showing absence of intracardiac thrombi.
7. Patients who have undergone a trans-esophageal echocardiogram within the last 48 hours.

Inclusion Criteria for the Phase II Component

1. Patients with spontaneous AF
2. Patients with or without structural Heart Disease.
3. Men or Women aged 18 years or older.
4. Patients undergoing an invasive catheterization procedure including right heart catheterization.
5. Patients who give an informed consent for participation in the study.
6. Patients who have undergone a trans-thoracic echocardiogram within the last 14 days showing absence of intracardiac thrombi.

Exclusion Criteria:

Exclusion Criteria for the Phase I Component

1. Patients in whom placement of an ICE catheter for adequate atrial visualization is technically not feasible.
2. Women of child bearing potential, in whom pregnancy cannot be excluded.
3. Patients with any medical condition or social circumstance, which in the opinion of the investigator, would make the patient's successful completion of the study doubtful

Exclusion Criteria for the Phase II Component 1. Patients anticoagulated for > 7 days. 2. Patients who have had a cardioembolic event within the last 1-month. 3. Patients requiring urgent cardioversion due to hemodynamic instability. 4. Patients in whom placement of an ICE catheter for adequate atrial visualization is technically not feasible. 5. Patients with contraindications for Warfarin. 6. Women of child bearing potential, in whom pregnancy cannot be excluded. 7. Patients who need anticoagulation withdrawn due to an elective procedure 8. Patients with any medical condition or social circumstance, which in the opinion of the investigator would make the patient's successful completion of the study doubtful.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2005-03; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of thrombi or spontaneous contrast detected by ICE or TEE | intraoperative
  Prevalence of thrombi or spontaneous contrast detected by ICE

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Saksena, MD, FACC, Study Chair — Professor, UMDNJ-RWJ Medical School
Locations (6):
- United States (5):
  - Mayo Clinic, Jacksonville, Florida
  - University of Chicago - Center for Advanced Medicine, Chicago, Illinois
  - Carle Clinic, Urbana, Illinois
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Aurora Sinai Medical Center / St. Lukes Medical Center, Milwaukee, Wisconsin
- Erasmus University Medical Center, Rotterdam, Rotterdam, Netherlands

REFERENCES:
- [Background] Pearson AC, Labovitz AJ, Tatineni S, Gomez CR. Superiority of transesophageal echocardiography in detecting cardiac source of embolism in patients with cerebral ischemia of uncertain etiology. J Am Coll Cardiol. 1991 Jan;17(1):66-72. doi: 10.1016/0735-1097(91)90705-e. PMID 1987242
- [Background] Lin SL, Hsu TL, Liou JY, Chen CH, Chang MS, Chiang HT, Chen CY. Usefulness of transesophageal echocardiography for the detection of left atrial thrombi in patients with rheumatic heart disease. Echocardiography. 1992 Mar;9(2):161-8. doi: 10.1111/j.1540-8175.1992.tb00454.x. PMID 10149880
- [Background] Castello R, Pearson AC, Labovitz AJ. Prevalence and clinical implications of atrial spontaneous contrast in patients undergoing transesophageal echocardiography. Am J Cardiol. 1990 May 1;65(16):1149-53. doi: 10.1016/0002-9149(90)90330-4. PMID 2330903
- [Background] Klein AL, Grimm RA, Murray RD, Apperson-Hansen C, Asinger RW, Black IW, Davidoff R, Erbel R, Halperin JL, Orsinelli DA, Porter TR, Stoddard MF; Assessment of Cardioversion Using Transesophageal Echocardiography Investigators. Use of transesophageal echocardiography to guide cardioversion in patients with atrial fibrillation. N Engl J Med. 2001 May 10;344(19):1411-20. doi: 10.1056/NEJM200105103441901. PMID 11346805
- [Background] Packer DL, Stevens CL, Curley MG, Bruce CJ, Miller FA, Khandheria BK, Oh JK, Sinak LJ, Seward JB. Intracardiac phased-array imaging: methods and initial clinical experience with high resolution, under blood visualization: initial experience with intracardiac phased-array ultrasound. J Am Coll Cardiol. 2002 Feb 6;39(3):509-16. doi: 10.1016/s0735-1097(01)01764-8. PMID 11823090
- [Background] Olgin JE, Kalman JM, Fitzpatrick AP, Lesh MD. Role of right atrial endocardial structures as barriers to conduction during human type I atrial flutter. Activation and entrainment mapping guided by intracardiac echocardiography. Circulation. 1995 Oct 1;92(7):1839-48. doi: 10.1161/01.cir.92.7.1839. PMID 7671368
- [Background] Epstein LM, Smith T, TenHoff H. Nonfluoroscopic transseptal catheterization: safety and efficacy of intracardiac echocardiographic guidance. J Cardiovasc Electrophysiol. 1998 Jun;9(6):625-30. doi: 10.1111/j.1540-8167.1998.tb00945.x. PMID 9654229
- [Background] Marrouche NF, Martin DO, Wazni O, Gillinov AM, Klein A, Bhargava M, Saad E, Bash D, Yamada H, Jaber W, Schweikert R, Tchou P, Abdul-Karim A, Saliba W, Natale A. Phased-array intracardiac echocardiography monitoring during pulmonary vein isolation in patients with atrial fibrillation: impact on outcome and complications. Circulation. 2003 Jun 3;107(21):2710-6. doi: 10.1161/01.CIR.0000070541.83326.15. Epub 2003 May 19. PMID 12756153
- [Background] Mudra H, Klauss V, Blasini R, Kroetz M, Rieber J, Regar E, Theisen K. Ultrasound guidance of Palmaz-Schatz intracoronary stenting with a combined intravascular ultrasound balloon catheter. Circulation. 1994 Sep;90(3):1252-61. doi: 10.1161/01.cir.90.3.1252. PMID 8087934
- [Background] Hijazi Z, Wang Z, Cao Q, Koenig P, Waight D, Lang R. Transcatheter closure of atrial septal defects and patent foramen ovale under intracardiac echocardiographic guidance: feasibility and comparison with transesophageal echocardiography. Catheter Cardiovasc Interv. 2001 Feb;52(2):194-9. doi: 10.1002/1522-726x(200102)52:23.0.co;2-4. PMID 11170327
- [Background] Ren JF, Marchlinski FE, Callans DJ. Left atrial thrombus associated with ablation for atrial fibrillation: identification with intracardiac echocardiography. J Am Coll Cardiol. 2004 May 19;43(10):1861-7. doi: 10.1016/j.jacc.2004.01.031. PMID 15145112
- [Background] Shanewise JS, Cheung AT, Aronson S, Stewart WJ, Weiss RL, Mark JB, Savage RM, Sears-Rogan P, Mathew JP, Quinones MA, Cahalan MK, Savino JS. ASE/SCA guidelines for performing a comprehensive intraoperative multiplane transesophageal echocardiography examination: recommendations of the American Society of Echocardiography Council for Intraoperative Echocardiography and the Society of Cardiovascular Anesthesiologists Task Force for Certification in Perioperative Transesophageal Echocardiography. J Am Soc Echocardiogr. 1999 Oct;12(10):884-900. doi: 10.1016/s0894-7317(99)70199-9. No abstract available. PMID 10511663
- [Background] Petersen P, Boysen G, Godtfredsen J, Andersen ED, Andersen B. Placebo-controlled, randomised trial of warfarin and aspirin for prevention of thromboembolic complications in chronic atrial fibrillation. The Copenhagen AFASAK study. Lancet. 1989 Jan 28;1(8631):175-9. doi: 10.1016/s0140-6736(89)91200-2. PMID 2563096
- [Background] Boston Area Anticoagulation Trial for Atrial Fibrillation Investigators; Singer DE, Hughes RA, Gress DR, Sheehan MA, Oertel LB, Maraventano SW, Blewett DR, Rosner B, Kistler JP. The effect of low-dose warfarin on the risk of stroke in patients with nonrheumatic atrial fibrillation. N Engl J Med. 1990 Nov 29;323(22):1505-11. doi: 10.1056/NEJM199011293232201. PMID 2233931
- [Background] Stroke Prevention in Atrial Fibrillation Study. Final results. Circulation. 1991 Aug;84(2):527-39. doi: 10.1161/01.cir.84.2.527. PMID 1860198
- [Background] Connolly SJ, Laupacis A, Gent M, Roberts RS, Cairns JA, Joyner C. Canadian Atrial Fibrillation Anticoagulation (CAFA) Study. J Am Coll Cardiol. 1991 Aug;18(2):349-55. doi: 10.1016/0735-1097(91)90585-w. PMID 1856403
- [Background] Secondary prevention in non-rheumatic atrial fibrillation after transient ischaemic attack or minor stroke. EAFT (European Atrial Fibrillation Trial) Study Group. Lancet. 1993 Nov 20;342(8882):1255-62. PMID 7901582
- [Background] Warfarin versus aspirin for prevention of thromboembolism in atrial fibrillation: Stroke Prevention in Atrial Fibrillation II Study. Lancet. 1994 Mar 19;343(8899):687-91. PMID 7907677
- [Background] Adjusted-dose warfarin versus low-intensity, fixed-dose warfarin plus aspirin for high-risk patients with atrial fibrillation: Stroke Prevention in Atrial Fibrillation III randomised clinical trial. Lancet. 1996 Sep 7;348(9028):633-8. PMID 8782752
- [Background] Petersen P, Grind M, Adler J; SPORTIF II Investigators. Ximelagatran versus warfarin for stroke prevention in patients with nonvalvular atrial fibrillation. SPORTIF II: a dose-guiding, tolerability, and safety study. J Am Coll Cardiol. 2003 May 7;41(9):1445-51. doi: 10.1016/s0735-1097(03)00255-9. PMID 12742279
- [Background] Olsson SB; Executive Steering Committee of the SPORTIF III Investigators. Stroke prevention with the oral direct thrombin inhibitor ximelagatran compared with warfarin in patients with non-valvular atrial fibrillation (SPORTIF III): randomised controlled trial. Lancet. 2003 Nov 22;362(9397):1691-8. doi: 10.1016/s0140-6736(03)14841-6. PMID 14643116
- [Background] Fuster V, Ryden LE, Asinger RW, Cannom DS, Crijns HJ, Frye RL, Halperin JL, Kay GN, Klein WW, Levy S, McNamara RL, Prystowsky EN, Wann LS, Wyse DG; American College of Cardiology; American Heart Association; European Society of Cardiology; North American Society of Pacing and Electrophysiology. ACC/AHA/ESC guidelines for the management of patients with atrial fibrillation. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines and Policy Conferences (Committee to develop guidelines for the management of patients with atrial fibrillation) developed in collaboration with the North American Society of Pacing and Electrophysiology. Eur Heart J. 2001 Oct;22(20):1852-923. doi: 10.1053/euhj.2001.2983. No abstract available. PMID 11601835
- [Derived] Saksena S, Sra J, Jordaens L, Kusumoto F, Knight B, Natale A, Kocheril A, Nanda NC, Nagarakanti R, Simon AM, Viggiano MA, Lokhandwala T, Chandler ML; ICE-CHIP Investigator Study Group. A prospective comparison of cardiac imaging using intracardiac echocardiography with transesophageal echocardiography in patients with atrial fibrillation: the intracardiac echocardiography guided cardioversion helps interventional procedures study. Circ Arrhythm Electrophysiol. 2010 Dec;3(6):571-7. doi: 10.1161/CIRCEP.110.936161. Epub 2010 Sep 18. PMID 20852299